CLINICAL TRIAL: NCT00389233
Title: A Randomised, Multi-Centre, Single-Blinded, Pivotal Phase III Trial to Assess the Efficacy, Acceptability and Safety of a New 2 Litre Gut Cleansing Solution NRL994 Versus a Standard Colon Preparation With 4L PEG+E.
Brief Title: A Phase III Trial to Assess the Efficacy, Acceptability and Safety of Moviprep® Versus a 4L PEG+E Standard Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Hans-Jürgen Gruss, Norgine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRL994-01/2001
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Colonoscopy
MeSH Terms: interventions — MoviPrep; klean prep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2L gut cleansing solution
  Interventions: Drug: Macrogol3350 NA sulphate NACl KCl ascorbic acid NA ascorbate
- 2 (Active Comparator): 4L preparation
  Interventions: Drug: Macrogol3350 Na sulphate Na bicarbonate NaCl KCl

INTERVENTIONS:
Drug: Macrogol3350 NA sulphate NACl KCl ascorbic acid NA ascorbate — 1 pack will consist of 2L NRL 994 - 4 (2 x PEG + E/"P" + 2 x Vitamin C/"C") sachets for the 2L of 2 sachets (1 x "P" plus 1 x "C") will be dissolved in 1L of water. Each litre will be drunk within 1 hour followed by at least 500ml of any additional clear fluid.
  Other Names: MOVIPREP®
  Arms: 1
Drug: Macrogol3350 Na sulphate Na bicarbonate NaCl KCl — 1 pack will consist of 4L PEG + E - contains 4 sachets for the 4L of PEG + E/"P/E". Each sachet will be dissolved in 1L of water. Each litre will be drunk within 1 hour.
  Other Names: KLEAN-PREP®
  Arms: 2

SUMMARY:
The study was carried out as a randomised, single-blind, active-controlled, multi-centric, phase III study with two parallel treatment groups. The primary efficacy criterion was the frequency of effective gut cleansing in each of the two treatment groups (grade A or B "overall quality of gut cleansing" as judged by a blinded expert panel on the basis of videotapes recorded during the endoscopic procedure).

DETAILED DESCRIPTION:
The study was designed as a randomised, active-controlled, single-blind, multi-centre, pivotal phase III trial with two parallel treatment groups. 15 German hospitals with specialised gastroenterology units were expected to participate in the investigation.

Up to 360 hospital in-patients routinely scheduled to undergo complete colonoscopy were to be enrolled one to two days prior to the endoscopic procedure, and to be randomly allocated to one of the two treatment arms in a ratio of 1:1. Bowel preparation was performed using equal split doses of either low-volume NRL994 (two doses of 1,000 mL each) or high-volume PEG+E (two doses of 2,000 mL each). The first dose was to be taken in the evening before the procedure, the second dose on the morning of the day of the colonoscopy. The patients allocated to NRL994 were asked to drink at least 1L of additional clear liquid in addition to the study drug. During colonoscopy the cleansing of each of the five pre-defined gut segments was to be assessed by the physician performing the examination, using a 5-level verbal rating scale. Videotapes were to be recorded of all procedures in order to allow central review by a blinded and independent expert panel whose ratings were the primary basis for the analysis of efficacy. The patients enrolled in the study were asked to fill in a questionnaire concerning the acceptability of the preparation. A patient's participation in the study was terminated upon completion of the intervention by performing a final examination and filling in the study termination page. No interim analysis was to be performed.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent prior to inclusion;
* male or female in-patients, aged 18 to 85 years, with indication for complete colonoscopy;
* willing and able to complete the entire procedure and to comply with study instructions;
* females of childbearing potential employing an adequate method of contraception.

Exclusion Criteria:

* ileus;
* intestinal obstruction or perforation;
* toxic megacolon;
* congestive heart failure (NYHA class III and IV);
* acute life-threatening cardiovascular disease;
* untreated or uncontrolled arterial hypertension (SBP max>170mmHg, DBP min>100mmHg);
* severe renal failure;
* severe liver failure;
* known glucose-6-phosphatase dehydrogenase deficiency;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2002-06; Study Completion 2002-12

PRIMARY OUTCOMES:
The frequency of effective gut cleansing in each of the two treatment groups (grade A or B "overall quality of gut cleansing" as judged by a blinded expert panel on the basis of videotapes recorded during the endoscopic procedure).

SECONDARY OUTCOMES:
Degree of gut cleansing in each of the five colonic segments
mean degree of gut cleansing
global quality of gut cleansing
overall ease to perform colonoscopy
degree of patient satisfaction
overall acceptability of the gut cleansing regimen
global taste evaluation of the solution,problems drinking the entire volume of gut cleansing solution
acceptability of the diet associated with the intake of the solution
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ell, Prof Dr med, Principal Investigator — Dept. of Internal Medicine II, Dr.-Horst-Schmidt Hospital, Teaching Hospital of the University Mainz
Locations (12):
- Germany (12):
  - Chefarzt der Abt. Gastroenterologie, Klinikum St. Marien, Amberg
  - Chefarzt Innere Medizin, Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Dachau, Innere Medizin - Gastroenterologie, Dachau
  - Chefarzt, Katholisches Krankenhaus St. Johann Nepomuk, Erfurt
  - Waldkrankenhaus St. Marien,, Erlangen
  - Zentrum für Innere Medizin,, Essen
  - Bürgerhospital Frankfurt e.V., Abteilung für interventionelle Endoskopie, Frankfurt am Main
  - Städtische Kliniken Frankfurt-Höchst, Frankfurt am Main
  - Klinikum Fürth, Med. Klinik II, Fürth
  - Abteilung für Innere Medizin, Israelitisches Krankenhaus, Hamburg
  - Kreiskrankenhaus, Tirschenreuth
  - Dr.-Horst-Schmidt-Kliniken GmbH, Innere Medizin II, Wiesbaden

REFERENCES:
- [Result] Ell C, Fischbach W, Bronisch JH, et al. Ergebnisse einer randomisierten, multizentrischen verblindeten Vergleichsstudie zur Wirksamkeit, Akzeptanz und Sicherheit einer neuen 2 Liter Darmvorbereitungslosung (Moviprep) im Vergleich zu einer etablierten 4 Liter Golytely Losung.[Results of a randomised, multi-centre, single-blinded trial to compare the efficacy, acceptability and safety of a new 2-litre gut cleansing solution versus a standard 4-litre PEG+E solution.] Z Gastroenterol 2004;42:P169
- [Result] Ell C, Gruss HJ.Results of a Randomised, Multi-Centre, Single-Blind Trial to Compare the Efficacy, Acceptability and Safety of a New 2-Litre Gut Cleansing Solution Versus a Standard 4-Litre PEG+E Solution.Gastrointest Endosc 2004;59(5):AB125
- [Derived] Ell C, Fischbach W, Bronisch HJ, Dertinger S, Layer P, Runzi M, Schneider T, Kachel G, Gruger J, Kollinger M, Nagell W, Goerg KJ, Wanitschke R, Gruss HJ. Randomized trial of low-volume PEG solution versus standard PEG + electrolytes for bowel cleansing before colonoscopy. Am J Gastroenterol. 2008 Apr;103(4):883-93. doi: 10.1111/j.1572-0241.2007.01708.x. Epub 2008 Jan 11. PMID 18190651